CLINICAL TRIAL: NCT00512395
Title: Influence of Epidural Analgesia in Elective Laparoscopic Colorectal Resections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Triemli Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STZ 13/04
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: laparoscopic colorectal surgery; epidural analgesia; pain score; postoperative ileus
MeSH Terms: conditions — Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): epidural analgesia
  Interventions: Drug: epidural analgesia (Duracain/Fentanyl/Naropin)
- 2 (No Intervention): traditional analgesia with opioids

INTERVENTIONS:
Drug: epidural analgesia (Duracain/Fentanyl/Naropin) — naropin 0.3% or duracain 0.125% + Fentanyl via epidural catheter 4-12 ml/h
  Arms: 1

SUMMARY:
Epidural anaesthesia in open surgery is a effective method for analgesia and has a positive effect on postoperative resolution of ileus. In laparoscopic surgery, the role of epidural surgery is not established. This prospective observational trial evaluates the effect of epidural analgesia in patients undergoing elective, laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
All patients with elective, laparoscopic colorectal resection between November 2004 and January 2007 were included in the trial. The decision for epidural analgesia was made by the anaesthetist and the patient. Contraindications were previous back surgery, coagulopathy, severe spondylarthrosis and refusal by the patient as contraindications.

Primary outcome was subjective feeling postoperatively, assessed with a VAS for pain and cramps and amount of analgesics used. Secondary outcomes were duration of postoperative bowel dismotility (first flatus, first defecation, first solid food intake) and general and specific morbidity.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic colorectal resection

Exclusion Criteria:

* emergency surgery
* preoperatively planned stoma formation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-11; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
pain (VAS), cramps (VAS) and quantity of analgesics | 8 days

SECONDARY OUTCOMES:
duration of postoperative ileus morbidity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Triemli Hospital, Zurich, Switzerland